CLINICAL TRIAL: NCT01980342
Title: Pharmacokinetics and Pharmacodynamics of the Etonogestrel Contraceptive Implant When Co-administered With Efavirenz
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: loss of funding
Sponsor: Johns Hopkins University (Other)
Collaborators: American College of Obstetricians and Gynecologists (Other); The Campbell Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NA_00087585
Record Dates: First submitted 2013-11-04; First posted 2013-11-08 (Estimated); Results first posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Drug Interaction
Keywords: Long acting reversible contraception; HIV
MeSH Terms: interventions — efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Efavirenz (Experimental): Healthy, reproductive-age women using the etonogestrel contraceptive implant who will take a two-week course of efavirenz 400 mg orally each night.
  Interventions: Drug: Efavirenz

INTERVENTIONS:
Drug: Efavirenz — Healthy women who are using Nexplanon will be asked to take a 2-week course of reduced-dose efavirenz (400 mg daily).
  Other Names: Sustiva

SUMMARY:
This study evaluates whether there is an interaction between etonogestrel, the progestin hormone released by the contraceptive implant Nexplanon, and efavirenz, a common medication used to treat HIV. The endpoints measured in this study will help determine if such an interaction leads to decreased contraceptive efficacy of the contraceptive implant.

DETAILED DESCRIPTION:
Women now make up nearly half of the world's HIV-infected population, and many of these women with HIV are of reproductive age. There is a growing need to provide effective contraception for those women who want or need to be protected against pregnancy. However, there is concern for decreased contraceptive efficacy in women on antiretroviral therapy who rely on hormonal contraception due to drug-drug interactions. Of particular concern is a possible interaction with etonogestrel, the active hormone in a long-acting reversible contraceptive implant. We propose a pilot study to evaluate the effect of efavirenz (EFV), a commonly used non-nucleoside reverse transcriptase inhibitor, on the pharmacokinetics of the etonogestrel implant. We will recruit 18 healthy women who have had the implant in place for 12 to 24 months. They will be asked to take a two-week course of efavirenz. During these two weeks and for four additional weeks, we will monitor semi-weekly etonogestrel concentrations, and serum, ultrasound, and cervical mucus markers of ovulation. We will also assess efavirenz concentration at baseline and at the end of the two-week treatment course. We will derive pharmacokinetic parameters and compare concentrations across time points. Results will help to inform the design of larger studies, and of similar studies with different antiretroviral medications. We hypothesize that taking efavirenz while using the etonogestrel contraceptive implant will not result in an increased incidence of ovulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women aged 18-40 years who have a Nexplanon®/Implanon® in place that is palpable on exam, had the device placed between 12 and 24 months prior to enrollment, and can provide documentation of when the implant was placed
* Able to speak and read English
* Documented HIV-negative status within 30 days of enrollment
* BMI between 18.5 and 24.9 kg/m2
* Willingness to take a two-week course of efavirenz
* Willingness to comply with study visit schedule (as described below), including blood sampling, transvaginal ultrasounds, and cervical mucus assessment
* Negative urine human chorionic gonadotropin pregnancy test at study entry
* Normal laboratory values within 30 days of study entry, as specified below:

  * White blood cell count ≥ 4500 and ≤ 11000 cells/mm3
  * Platelet count ≥ 100,000 platelets/mm3
  * Hemoglobin ≥ 8.0 g/dL
  * International normalized ratio (INR) ≤ 1.8
  * Aspartate transaminase (SGOT) and alanine aminotransferase (SGPT) ≤ 3 times the upper limit of normal (ULN) (upper limit of normal)
  * Creatinine ≤ 1.5 x ULN
  * Serum amylase ≤ 1.5 x ULN
  * Total bilirubin ≤ 2.0 x ULN
* Agree to use an additional reliable method of contraception while participating in the study. Acceptable methods include:

  * Abstinence
  * Condoms (male or female) with or without spermicide
  * Pre-existing sterilization of subject or her male partner
* Willingness to abstain from alcohol consumption during the study period
* Willingness to abstain from any grapefruit product or supplement for the duration of the study.

Exclusion Criteria:

* Breastfeeding
* Hypersensitivity to efavirenz
* History of seizure disorder
* Initiated, discontinued, or changed doses of drugs that are cytochrome P450 isoenzyme 3A4 (CYP3A4) inducers or inhibitors within 30 days of study entry.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2014-10; Primary Completion 2018-04-04 (Actual); Study Completion 2018-04-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins University Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Efavirenz
Started | 1
Completed | 0
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Efavirenz
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Serum Concentration of Etonogestrel Before and After Two Weeks of Efavirenz
Description: We will draw a baseline serum etonogestrel immediately prior to a participant starting the 2-week course of efavirenz. Serial blood samples will subsequently be drawn over the next 6 weeks to assess for changes in serum etonogestrel concentration. We will be looking to see if the serum etonogestrel concentration decreases below the level necessary for reliable ovulation suppression.
Time Frame: 6 weeks
Population: No data was collected for this outcome measure as the study was terminated prematurely after enrolling only 1 participant.
Arm/Group | Efavirenz
Number analyzed (Participants) | 0

2. Secondary Outcome: Serum Efavirenz Concentrations at the Start and End of the 2-week Dosing Period
Description: We will assess serum efavirenz concentrations at the beginning and end of the 2-week dosing period. By comparing these concentrations to historical controls, we will determine whether taking efavirenz while using the etonogestrel implant alters the serum concentration of efavirenz.
Time Frame: 2 weeks
Population: as for outcome 1
Arm/Group | Efavirenz
Number analyzed (Participants) | 0

3. Secondary Outcome: Serum Hormone Markers of Ovulation
Description: We will test serial blood samples for levels of luteinizing hormone (LH), follicle stimulating hormone (FSH), estradiol, and progesterone to determine whether the etonogestrel implant is able to suppress ovulation during and after a course of efavirenz.
Time Frame: 6 weeks
Population: as for outcome 1
Arm/Group | Efavirenz
Number analyzed (Participants) | 0

4. Secondary Outcome: Transvaginal Ultrasound to Assess for Ovarian Follicular Development
Description: For the entire 6 week period of the study, participants will undergo twice-weekly transvaginal ultrasound to assess for the development of ovarian follicles. This direct assessment of follicular development will be combined with serum hormone concentrations to determine if efavirenz increases the incidence of ovulation in women using the etonogestrel implant for contraception.
Time Frame: 6 weeks
Population: as for outcome 1
Arm/Group | Efavirenz
Number analyzed (Participants) | 0

5. Secondary Outcome: Cervical Mucus Quality
Description: Cervical mucus quality will be assessed twice weekly throughout the study period. The etonogestrel implant exerts a secondary contraceptive effect by causing cervical mucus to become thick and sticky, and therefore less permissive to the movement of sperm through the female genital tract. We will assess whether efavirenz causes a change in cervical mucus quality that would make sperm penetration more likely, and therefore indicate a reduction in the implant's contraceptive effect.
Time Frame: 6 weeks
Population: as for outcome 1
Arm/Group | Efavirenz
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Data was not collected due to study termination
Description: This study was terminated early due to loss of funding. There was only 1 participant enrolled. No Adverse Event Data was collected
Arm/Group | Efavirenz
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-05): https://cdn.clinicaltrials.gov/large-docs/42/NCT01980342/Prot_SAP_000.pdf